CLINICAL TRIAL: NCT02021708
Title: Effect of Shisha Smoking on the Biology of the Airway Epithelium in Qatar
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Weill Cornell Medical College in Qatar (Other); Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-00055 [JIRB]; NPRP 09-742-3-194 (Other: Qatar National Research Fund)
Record Dates: First submitted 2013-11-22; First posted 2013-12-27 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Non-smoker: This group will include individuals without any history of lung disease, including asthma, and without recurrent or acute pulmonary disease. Individuals must also have smoked less than 100 cigarettes and/or less than 10 shisha pipes in their lifetime.
- Shisha smoker: This group will include individuals who have a shisha smoking history of more than 5 pipe-years and must currently smoke more than 5 pipes per week. Individuals must not show any signs of acute lung infection or have medical history of significant illness or other significant medical issues.
- Cigarette smoker: This group will include individuals who have a cigarette smoking history that will be confirmed by urine testing. Individuals must not show any signs of acute lung infection or have medical history of significant illness or other significant medical issues.

SUMMARY:
The purpose of this study is to learn about the effects of smoking shisha on the lungs, when compared to the effects of smoking cigarettes or of not smoking. The investigators hope to learn more about how shisha smokers should be monitored and treated once diseased.

DETAILED DESCRIPTION:
Traditional shisha smoking is practiced by ~10% of the Qatari adult population. Although based on tobacco leaves, shisha smoking exposes the airway epithelium to a chemical insult of intensity and duration different from that of cigarette smoking. This study, a collaboration between WCMC-Qatar and WCMC-New York and the Hamad Medical Corporation (HMC), is focused on defining the biology of the airway epithelium of shisha smokers compared to non-smokers. Using approved protocols, bronchoscopy will be used to sample the airway epithelium, the site of the earliest changes associated with smoking. The transcriptome of the recovered epithelium will be assessed in the genomic core WCMC-Qatar for gene expression using microarrays and complete RNA sequencing using massive parallel sequencing.Based on this information, the epithelial DNA will be assessed for relevant SNPs, copy number variations and methylation status. Parallel studies will be carried out in cigarette smokers, providing a comprehensive catalog of shisha smoking-induced changes compared to cigarette smokers and non-smokers in this population.

ELIGIBILITY:
Non-smoker

Inclusion Criteria:

* Population living in Qatar
* Must provide informed consent
* Individuals must also have smoked less than 100 cigarettes and/or less than 10 shisha pipes in their lifetime
* Has normal pulmonary function test
* Has normal chest xray
* No signs of acute lung infection

Exclusion Criteria:

* Medical history of significant illness or other significant medical issues
* Regular shisha smoker
* Regular cigarette smoker
* Simultaneous cigarette plus shisha smoking

Shisha smoker

Inclusion Criteria:

* Population living in Qatar
* Must provide informed consent
* Must have smoked 5 pipe-yr
* Must currently smoke 5 pipes/wk
* Has normal function tests
* Has normal chest xray
* No signs of acute lung infection

Exclusion Criteria:

* Medical history of significant illness or other significant medical issues
* Regular cigarette smoker
* Simultaneous cigarette plus shisha smoking

Cigarette smoker

Inclusion Criteria:

* Population living in Qatar
* Must provide informed consent
* Confirmation of smoking status by urine testing
* Confirmation of smoking status by assessment of carboxyhemoglobin
* Has normal function tests
* Has normal chest xray
* No signs of acute lung infection

Exclusion Criteria:

* Medical history of significant illness or other significant medical issues
* Regular shisha smoker
* Simultaneous cigarette plus shisha smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited in the pulmonary and smoking cessation clinics of HMC.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Gene expression changes in the small airway epithelium (SAE) | 3 days
  We will measure the effect that shisha smoking has on the small airway epithelium (SAE) by measuring parameters such as the SAE gene expression in shisha smokers (i.e., non-cigarette smokers). We will compare these parameters to the same parameters measured in non-smokers and cigarette smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Walters, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided